CLINICAL TRIAL: NCT04411069
Title: Simplified Algorithm for the Prevention of Postoperative Nausea and Vomiting in an Oncological Hospital
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NP 1336/18
Record Dates: First submitted 2020-05-18; First posted 2020-06-02 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Nausea; Postoperative Vomiting
Keywords: nausea; vomiting; chemoterapy
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Droperidol

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient didn't know if he received the third anti emetic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients without previous CINV (No Intervention): Patients who didn't have chemotherapy or that didn´t have any nausea and/or vomiting induced by chemotherapy (CINV) before surgery
- Patients with previous CINV (Other): Patients who had previous nausea and vomiting induced by chemoterapy.
  Interventions: Drug: Droperidol

INTERVENTIONS:
Drug: Droperidol — Pacients who had nausea and vomiting induced by chemotherapy will receive three anti emetic drugs: 4mg dexametasone, 4 mg ondansetron and 0,625 mg droperidol
  Other Names: Intravenous droperidol
  Arms: Patients with previous CINV

SUMMARY:
Previous history of nausea and vomiting induced by prior chemotherapy still not included as predictive factor of postoperative nausea and vomiting, although has been demonstrated that has influence in postoperative outcome.

The project aims to evaluate the efficacy of a simplified algorithm in prevention postoperative nausea and vomiting , with pacients with previous history of nausea and vomiting induced by prior chemotherapy, submitted to medium or large surgery.

DETAILED DESCRIPTION:
Quasi-experimental study, with evaluation after the application of a specific postoperative nausea and vomiting prevention algorithm for cancer patients.

The study will be carried out in 2 phases:

Phase 1: Team training. In this phase, a protocol was established for PONV prophylaxis, using two questions:

1. Patient undergoing chemotherapy before surgery;
2. Patient presented chemotherapy induced nausea and vomiting (CINV).

If the answer is yes to both questions, the anesthetist administers 3 antiemetics (4mg dexametasone, 4mg ondansetron and 0,625mg droperidol). If the answer is no to one of the questions, the anesthetist administers 2 antiemetics (4mg dexametasone and 4mg ondansetron); In this phase, educational measures will be implemented by team meetings and individual approach of all anesthesiologists at ICESP to present the study project and the algorithm. A summary of the the study will be sent daily through the social network Whats App®.

The number of patients was calculated taking into account adherence to the new prophylaxis protocol for post-operative nausea and vomiting. If we consider an alpha error of 5% and test power of 80%, to have a NVPO reduction of 41% (current overall incidence) to 25% (incidence after protocol adherence) in high-risk patients, we need to study 270 patients (135 each group adherence and non-adherence to the protocol).

Phase 2: Post-training assessment. In the second phase of the study, after the end of the dissemination of the protocol among doctors, the patients will be evaluated on the first postoperative day. The following variables were analyzed: sex, race, age, body mass index, general state of American Society of Anesthesiologist, Apfel scale, type of surgery and anesthesia, use and type of opioids, history of chemotherapy induced nausea and vomiting, type of antiemetics used in the operating room and in the first postoperative day, duration of anesthesia and surgery and nausea and vomiting in 6 and 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent medium to large surgery

Exclusion Criteria:

* Patients who are unable to communicate (orotracheal intubation after the surgery, confusion or agitation) or understand the Portuguese language;
* Insulin dependent patients
* Patients who underwent emergency surgery and neurosurgery
* Pacients who had an increased QT interval on the electrocardiogram
* History of allergy to dexametasone, ondansetron or droperidol
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | from 0 to 24 postoperative hours
  record of any episode of nausea and or vomiting in the 24 postoperative hours

SECONDARY OUTCOMES:
Changing in the institutional protocol | from the begining to the study to the end of the study (2 years)
  number of patients with chemotherapy-induced nausea and vomiting that received 3 antiemetics in the operating room

CONTACTS AND LOCATIONS:
Overall Officials: Roger Chammas, Study Director — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Cancer Institute of the State of Sao Paulo - ICESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No